CLINICAL TRIAL: NCT00480337
Title: In Vitro Maturation of Immature Oocytes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4317-AH-CTIL
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome
Keywords: PCOS; Fertility Preservation; Repeated IVF Failure; S/P Hyperstimulation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: In Vitro Maturation of immature oocytes

SUMMARY:
The aim of this study is to aspirate immature oocytes from antral follicles and mature the oocytes in vitro. These mature oocytes will serve for fertilization and the creation of embryos which will be replace in the uterus as performed during normal IVF.We will record the efficacy and safety of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS
* Women with previous Hyperstimulation or with risk of developing hyperstimulation during IVF Treatment
* Women diagnosed with cancer who are interested in fertility preservation
* Women with repeated IVF failure

Exclusion Criteria:

* Severe cases of endometriosis
* Large myomas
* Hydrosalpinxs Technical problem with previous oocytes pick-up

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Hourvitz, Principal Investigator — IVF Unit, Sheba Medical Center
Locations (1):
- IVF Unit, Shea Medical Center, Tel-Hashomer, Ramat Gan, Israel